CLINICAL TRIAL: NCT05700006
Title: An Observational Study of Women With Breast Cancer Examining the Effect of Endocrine Therapy on Aging
Brief Title: Pilot Observational Study Examining the Effect of Endocrine Therapy on Aging
Acronym: BETA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, N. Lynn Henry, Professor, University of Michigan
Other Study IDs: HUM00208684; UMCC 2021.129 (Other: Rogel Cancer Center)
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasm Female; Arthralgia; Aging
Keywords: aromatase inhibitor; microbiome
MeSH Terms: conditions — Arthralgia | interventions — Aromatase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Age 65+, AI therapy: Postmenopausal women age 65 and older who are starting treatment with standard of care aromatase inhibitor therapy
  Interventions: Drug: Aromatase inhibitor
- Age 65+, no endocrine therapy: Postmenopausal women age 65 and older who are not starting treatment with any endocrine therapy
- Age under 65, AI therapy: Postmenopausal women age less than 65 who are starting treatment with standard of care aromatase inhibitor therapy
  Interventions: Drug: Aromatase inhibitor

INTERVENTIONS:
Drug: Aromatase inhibitor — Standard of care anastrozole, exemestane, or letrozole
  Groups: Age 65+, AI therapy; Age under 65, AI therapy

SUMMARY:
The goal of this pilot observational study is to learn about the feasibility of collecting patient-reported data and stool and blood samples from patients age 65 and older treated with aromatase inhibitor therapy for breast cancer. Participants will be treated with standard of care aromatase inhibitor therapy and will undergo serial phlebotomy, complete patient-reported questionnaires, and submit serial stool samples.

The main exploratory translational questions it aims to obtain preliminary data for are:

* What are the effects of aromatase inhibitor therapy on biomarkers of aging?
* What are the effects of aromatase inhibitor therapy on the microbiome? These data will be used for the development of future definitive studies.

ELIGIBILITY:
Inclusion Criteria

* Female gender.
* Cohort 1: Age 65 or greater. Cohort 2: Age younger than 65 years
* Cohort 1 Participants (starting AI therapy): Histologically proven stage 0-III carcinoma of the breast or at high risk for development of breast cancer who are planning to undergo treatment with neoadjuvant or adjuvant aromatase inhibitor therapy (anastrozole, letrozole, or exemestane).
* Cohort 1 Controls (no endocrine therapy): Histologically proven stage 0-III carcinoma of the breast or high risk for development of breast cancer and who are not planning to undergo treatment with any endocrine therapy (AI or tamoxifen).
* Participants Cohort 2 (starting AI therapy): Histologically proven stage 0-III carcinoma of the breast or at high risk for development of breast cancer who are planning to undergo treatment with neoadjuvant or adjuvant aromatase inhibitor therapy (anastrozole, letrozole, or exemestane).
* Concurrent treatment with GnRHa therapy, radiation therapy, CDK4/6 inhibitor, bisphosphonate, PARP inhibitor, and/or anti-HER2 therapy is permitted. Prior tamoxifen is permitted.
* The patient is aware of the nature of her diagnosis, understands the study requirements, risks, and discomforts, and is able and willing to sign an informed consent form.
* Able to read and understand English.

Exclusion Criteria

* Distant metastatic disease
* Prior aromatase inhibitor therapy except in the context of fertility treatment.
* Use of exogenous estrogen supplementation other than vaginal estrogen preparations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer or who are at high risk for breast cancer who are starting treatment with aromatase inhibitor therapy as standard of care for treating breast cancer or for chemoprevention will be eligible. In addition, women age 65 and older with breast cancer or at high risk for developing breast cancer who are not going to receive treatment with endocrine therapy are eligible for the control cohort.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of particpants in the 65+ AI therapy group who complete 3 serial blood collections and 5 serial ePRO collections | 1 year
  To assess feasibility of enrolling patients 65 and older in a study that collects serial blood samples and electronic patient-reported outcomes

SECONDARY OUTCOMES:
Percentage of participants who submit at least 2 out of 3 requested serial stool samples | 12 weeks
  To assess feasibility of enrolling patients with breast cancer in a study that collects serial stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No